CLINICAL TRIAL: NCT05242211
Title: Protocols Adjustments for Cardio-Pulmonary Exercise Testing in Healthy Population
Brief Title: Cardio-Pulmonary Exercise Testing in Healthy Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Gur Mainzer, Head of the pediatric cardiology department, The Baruch Padeh Medical Center, Poriya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0020-17-POR
Record Dates: First submitted 2021-12-19; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Healthy Obesity, Metabolically
Keywords: exercise; maximal exercise test; exercise protocol; metabolic
MeSH Terms: conditions — Obesity, Metabolically Benign; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Healthy volunteers (normal and overweight ) will be recruited to participants in the study. Demographics (age, sex), anthropometric (height, weight, abdominal circumference), will be measured. By using questionnaire, physical activity behavior and motivation toward engage in physical activity will be filled by the participants. Each participants will conducted an exercise test on treadmill (using Modified Bruce Protocol) and cycle ergometer. Quark CPET metabolic cart (Cosmed, Rome, Italy) will be used to collect and analysis gas exchange. 10 minute after the graded exercise test Supra maximal exercise test (SMT) will be done for 2 minutes one stage (treadmill protocol) or 10% at cycle protocol higher than highest load achieved in the incremental test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy (Other): Healthy participants will do both cycle ergometer and treadmill exercise
  Interventions: Other: exercise test

INTERVENTIONS:
Other: exercise test — Each participants will conducted an exercise test on treadmill (using Modified Bruce Protocol) and cycle ergometer. Quark CPET metabolic cart (Cosmed, Rome, Italy) will be used to collect and analysis gas exchange. 10 minute after the graded exercise test Supra maximal exercise test (SMT) will be done for 2 minutes one stage (treadmill protocol) or 10% at cycle protocol higher than highest load achieved in the incremental test.

SUMMARY:
Introduction: Cardiopulmonary exercise test (CPET) is a helpful tool for evaluation of aerobic exercise capacity and tolerance for variety of population. The test progression include an incremental stepwise or ramp control protocol to exhaustion There are different methods used in various clinical setting. CPET involves the measurement of respiratory gas exchange i.e. oxygen uptake, carbon dioxide, minute ventilation, other variables while monitoring ECG, blood pressure, pulse oximetry and exertion perceived (Borg Scale) during an incremental test on a cycle-ergo meter or treadmill. This test allow to assess an integrative exercise responses to submaximal and maximal effort.

Aim: To compere exercise responses and achieved criteria for maximal exercise testing with different exercise protocol Methods: Healthy volunteers (normal and overweight ) will be recruited to participants in the study. Demographics (age, sex), anthropometric (height, weight, abdominal circumference), will be measured. By using questionnaire, physical activity behavior and motivation toward engage in physical activity will be filled by the participants. Each participants will conducted an exercise test on treadmill (using Modified Bruce Protocol) and cycle ergometer. Quark CPET metabolic cart (Cosmed, Rome, Italy) will be used to collect and analysis gas exchange. 10 minute after the graded exercise test Supra maximal exercise test (SMT) will be done for 2 minutes one stage (treadmill protocol) or 10% at cycle protocol higher than highest load achieved in the incremental test.

All exercise parameter done on the different ergometer will be compared

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-55

Exclusion Criteria:

* Physical activity limitation due to orthopedic , neurological and cognition deficit Pregnancy children

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-03 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
VO2 MAX | through study completion, an average of 1 year
  maximal oxygen consumption
RPE-rate of perceived exertion | through study completion, an average of 1 year
  rate of perceived exertion on a 10 point modified Borg scale
Max heart rate | through study completion, an average of 1 year
  Max heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Gur Mainzer, MD, Principal Investigator — The Baruch Padeh Medical Center, Poriya
Locations (1):
- The BARUCH PADEH Medical Center, Poriya, Tiberias, The Lower Galilee, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astorino TA, White AC, Dalleck LC. Supramaximal testing to confirm attainment of VO2max in sedentary men and women. Int J Sports Med. 2009 Apr;30(4):279-84. doi: 10.1055/s-0028-1104588. Epub 2009 Feb 6. PMID 19199208
- [Background] Bhammar DM, Stickford JL, Bernhardt V, Babb TG. Verification of Maximal Oxygen Uptake in Obese and Nonobese Children. Med Sci Sports Exerc. 2017 Apr;49(4):702-710. doi: 10.1249/MSS.0000000000001170. PMID 27875494
- [Background] Kaminsky LA, Whaley MH. Evaluation of a new standardized ramp protocol: the BSU/Bruce Ramp protocol. J Cardiopulm Rehabil. 1998 Nov-Dec;18(6):438-44. doi: 10.1097/00008483-199811000-00006. PMID 9857276
- [Background] Hawkins MN, Raven PB, Snell PG, Stray-Gundersen J, Levine BD. Maximal oxygen uptake as a parametric measure of cardiorespiratory capacity. Med Sci Sports Exerc. 2007 Jan;39(1):103-7. doi: 10.1249/01.mss.0000241641.75101.64. PMID 17218891
- [Background] Midgley AW, Carroll S, Marchant D, McNaughton LR, Siegler J. Evaluation of true maximal oxygen uptake based on a novel set of standardized criteria. Appl Physiol Nutr Metab. 2009 Apr;34(2):115-23. doi: 10.1139/H08-146. PMID 19370041
- [Background] Schaun GZ. The Maximal Oxygen Uptake Verification Phase: a Light at the End of the Tunnel? Sports Med Open. 2017 Dec 8;3(1):44. doi: 10.1186/s40798-017-0112-1. PMID 29218470
- [Background] Lafortuna CL, Lazzer S, Agosti F, Busti C, Galli R, Mazzilli G, Sartorio A. Metabolic responses to submaximal treadmill walking and cycle ergometer pedalling in obese adolescents. Scand J Med Sci Sports. 2010 Aug;20(4):630-7. doi: 10.1111/j.1600-0838.2009.00975.x. Epub 2009 Aug 23. PMID 19706003
- [Background] Mezzani A. Cardiopulmonary Exercise Testing: Basics of Methodology and Measurements. Ann Am Thorac Soc. 2017 Jul;14(Supplement_1):S3-S11. doi: 10.1513/AnnalsATS.201612-997FR. PMID 28510504
- [Background] Lollgen H, Leyk D. Exercise Testing in Sports Medicine. Dtsch Arztebl Int. 2018 Jun 15;115(24):409-416. doi: 10.3238/arztebl.2018.0409. PMID 29968559